CLINICAL TRIAL: NCT00220051
Title: A Phase II Study of Oxaliplatin (Eloxatin) Capecitabine (Xeloda) and Pre-operative Radiotherapy for Patients With Locally Advanced and Inoperable Rectal Cancer.
Brief Title: A Phase II Study of Oxaliplatin Capecitabine and Pre-operative Radiotherapy for Patients With Locally Advanced and Inoperable Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1973
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxaliplatin, Capecitabine
Procedure: Pre operative radiotherapy
Procedure: Surgical Resection

SUMMARY:
To assess the efficacy and safety of pre-operative capecitabine and oxaliplatin followed by capecitabine with concurrent radiotherapy followed by post-operative capecitabine in the treatment of patients with locally advanced or inoperable rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18.
* Histological diagnosis of adenocarcinoma of rectum.
* Locally advanced/ poor prognosis primary rectal cancer defined by MRI criteria of any of the categories below;

  * Tumour within 2 mm of mesorectal fascia ie circumferential resection margin threatened
  * Any T3 tumour at/below levatores
  * T3c tumour at any other level ie tumour extends >5 mm into peri-rectal fat
  * T4 tumour
  * Any T stage with 4 or more involved lymph nodes
* WHO performance status 0, 1 or 2.
* No evidence of metastatic disease as determined by CT scan of chest, abdomen, pelvis or other investigations such as PET scan or biopsy if required.
* Adequate bone marrow function with platelets > 100 X 109/l; WBC > 3 X 109/l; neutrophils > 1.5 X 109/l
* Normal renal function, with serum creatinine within the normal range or calculated creatinine clearance >50 ml/min.
* Adequate hepatic function with serum total bilirubin < 1.5 X upper limit of normal range.
* No concurrent uncontrolled medical conditions
* No previous malignant disease other than non-melanotic skin cancer or carcinoma in situ of the uterine cervix
* Adequate contraceptive precautions if relevant
* Informed written consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Presence of metastatic disease or recurrent rectal tumour
* Renal impairment (creatinine clearance<30 ml/min)
* Pregnancy or breast feeding
* Patients with a lack of physical integrity of the upper gastrointestinal tract, or known malabsorption syndromes
* Participation in any investigational drug study within the previous 4 weeks.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia even if controlled with medication) or myocardial infarction within the last 12 months)
* Patients with any symptoms or history of peripheral neuropathy.
* Prior pelvic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2001-11

PRIMARY OUTCOMES:
Pathological complete response rate.
Acute toxicity has been evaluated in previous phase I studies and should occur to a similar extent.

SECONDARY OUTCOMES:
Progression-free survival
Treatment related toxicity
Overall survival
Radiological response rate
Proportion of patients achieving pathological down staging compared with the pre-treatment MRI scan
Surgical complications
Bowel function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: D Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust

REFERENCES:
- [Derived] Chua YJ, Barbachano Y, Cunningham D, Oates JR, Brown G, Wotherspoon A, Tait D, Massey A, Tebbutt NC, Chau I. Neoadjuvant capecitabine and oxaliplatin before chemoradiotherapy and total mesorectal excision in MRI-defined poor-risk rectal cancer: a phase 2 trial. Lancet Oncol. 2010 Mar;11(3):241-8. doi: 10.1016/S1470-2045(09)70381-X. Epub 2010 Jan 25. PMID 20106720